CLINICAL TRIAL: NCT04593329
Title: National, Multicenter, Randomized, Double-blind, Triple-dummy, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Tiradentes Association in the Treatment of Acute Pain
Brief Title: Efficacy and Safety of Tiradentes Association in the Treatment of Acute Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategy review
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1519 - TIRADENTES 500/50
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Acute Pain
Keywords: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Dipyrone; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TIRADENTES (Experimental): The study is triple-dummy. The patient must take 3 pills, with a minimum interval of 6/6 hours for 3 days, if pain, as follows:
  1 tablet Tiradentes association, oral;
  1 capsule tramadol placebo, oral;
  1 tablet dipyrone placebo, oral.
  Interventions: Drug: TIRADENTES ASSOCIATION; Other: DIPYRONE PLACEBO; Other: TRAMADOL PLACEBO
- DIPYRONE (Active Comparator): The patient must take 3 pills, with a minimum interval of 6/6 hours for 3 days, if pain, as follows:
  1 tablet dipyrone, oral;
  1 tablet Tiradentes association placebo, oral;
  1 capsule tramadol placebo, oral.
  Interventions: Drug: DIPYRONE; Other: TIRADENTES ASSOCIATION PLACEBO; Other: TRAMADOL PLACEBO
- TRAMADOL (Active Comparator): The patient must take 3 pills, with a minimum interval of 6/6 hours for 3 days, if pain, as follows:
  1 capsule tramadol, oral;
  1 tablet dipyrone placebo, oral;
  1 tablet Tiradentes association placebo, oral.
  Interventions: Drug: TRAMADOL; Other: TIRADENTES ASSOCIATION PLACEBO; Other: DIPYRONE PLACEBO

INTERVENTIONS:
Drug: TIRADENTES ASSOCIATION — Tiradentes association tablet
  Arms: TIRADENTES
Drug: DIPYRONE — Dipyrone 500 mg
  Arms: DIPYRONE
Drug: TRAMADOL — Tramadol 50 mg
  Arms: TRAMADOL
Other: TIRADENTES ASSOCIATION PLACEBO — Tiradentes association placebo tablet
  Arms: DIPYRONE; TRAMADOL
Other: DIPYRONE PLACEBO — Dipyrone placebo tablet
  Arms: TIRADENTES; TRAMADOL
Other: TRAMADOL PLACEBO — Tramadol placebo capsule
  Arms: DIPYRONE; TIRADENTES

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Tiradentes association in adolescents and adults with acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Participants of both sexes, aged 15 years or more;
* Participants who require extraction of impacted mandibular third molar;
* Third molar with bone impactions observed in panoramic radiography, with classification of Winter (1926) mesioangular or vertical, and classification according to Pell & Gregory (1933) class II position B or class III position A or B;
* Participants with acute pain of moderate or severe intensity after completion of surgery.

Exclusion Criteria:

* Known hypersensitivity to the formula components used during the clinical trial;
* History of alcohol and/or substance abuse within 2 years;
* Participants whose surgery for molar extraction lasted more than 50 minutes;
* Participants with known gastroduodenal ulcers or diagnosis of persistent gastritis;
* Participants who used sedatives or hypnotic agents before surgery;
* Anesthesia technical failure or need for more than three anesthetic tubes;
* Participants with temporomandibular joint dysfunction or limited mouth opening;
* Surgical accident that, in the investigator's opinion, may interfere with the procedures or evaluations of the trial;
* Postoperative complications such as, but not restricted to: neuropraxia and paresthesia;
* Participants who used any medication that acts on the pain mechanism in the 3 days prior to the start of the trial;
* Participants under chronic opioid treatment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time-weighted Sum of Pain Intensity Difference Over 6 Hours (SPID0-6) | 0-6 hours
  Sum of pain intensity differences after 6 hours (SPID0-6), calculated as the weighted sum of pain intensity scale over 6 hours after the dose. Scoring is derived from the 4-point scale, which 0= no pain, 1= mild pain, 2= moderate pain and 4= severe pain.

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 26 days